CLINICAL TRIAL: NCT04067414
Title: A Single Cohort, Open-label, Multicenter, Dose-escalation Study of Safety and Efficacy of BZ019 for Adult CD19 Positive Relapsed and Refractory B-cell Non-Hodgkin Lymphoma
Brief Title: Exploratory Study of CD19-targeted Chimeric Antigen Receptor T Cells(BZ019) for Relapsed and Refractory B-cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Shanghai Cell Therapy Engineering Technology Research Center Group Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QT2018002
Record Dates: First submitted 2019-01-07; First posted 2019-08-26 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2024-05

CONDITIONS: Diffuse Large B Cell Lymphoma; High-grade B-cell Lymphoma; Transformed Lymphoma; Primary Mediastinal Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Intervention Model Description: A treatment program will include lymphodepleting chemotherapy with fludarabine and cyclophosphamide (flu/cy) followed by single-dose of BZ019 administered intravenously (IV). A 3×3 dose escalation design of BZ019 will be adopted.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BZ019 treatment (Experimental): Subjects will receive lymphodepleting chemotherapy of fludarabine and cyclophosphamide (flu/cy) followed by single-dose of BZ019 infusion. A 3×3 dose escalation design of BZ019 will be adopted.
  Interventions: Biological: BZ019

INTERVENTIONS:
Biological: BZ019 — Subjects will be enrolled in three dose-groups:
  Dose 1: 1×10^6/kg CAR+ cells; Dose 2: 3×10^6/kg CAR+ cells; Dose 3: 6×10^6/kg CAR+ cells.

SUMMARY:
This is an open-label, multicenter, dose-escalation phase 1 study to determine the safety and efficacy of BZ019 in relapsed or refractory CD19+ B-cell Lymphoma.

DETAILED DESCRIPTION:
This is an open-label, multicenter, phase 1 study to determine the safety and antitumor activity of BZ019 in adult patients with R/R large B cell lymphoma (DLBCL),including: DLBCL, not otherwise specified (NOS), transformed DLBCL, high-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements and primary mediastinal B-cell lymphoma (PMBCL).The safety and efficacy of a single dose of different target doses of BZ019 will be evaluated in the dose-escalation phase and dose-expansion phase.

Upon enrollment, subjects will undergo leukapheresis to enable BZ019 product generation. A baseline tumor biopsy (in subjects with accessible disease) and bone marrow aspirate and biopsy will be obtained.

Upon successful BZ019 product generation, subjects will enter the treatment phase and receive BZ019 infusion. A completed treatment program will include lymphodepleting chemotherapy with fludarabine and cyclophosphamide (flu/cy) followed by single-dose of BZ019 infusion. BZ019 will be administered 2 to 14 days after the completion of lymphodepleting chemotherapy.

After the infusion of BZ019, subjects will be in the follow-up period upon 12 months for evaluation the safety and efficacy of BZ019. Subjects will be followed for long-term safety, overall survival even after disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained prior to any screening procedures
2. Age ≥ 18 years subjects with Relapsed or refractory large B-cell lymphoma, including: DLBCL,NOS, high-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements, transformed B-cell lymphoma, primary mediastinal B-cell lymphoma (PMBCL).

   * No response for the last chemotherapy:

     * Progressive disease after the last chemotherapy or
     * Stable disease after the last chemotherapy, and the maintenance time for stable disease was no longer than 6 month after last dose.
   * Either having failed autologous Hematopoietic stem cell transplantation (ASCT), or being ineligible for or not consenting to ASCT

     * Refractory disease after ASCT or relapsed disease within 12 months after last ASCT (histologically confirmed) or
     * No response or relapsed disease for the last therapy after ASCT.
3. Subjects must be accepted adequate treatment, including at least:

   * Treated by CD20 monoclonal antibody (Rituximab) except for CD20 negative.
   * Chemotherapy including anthracycline
4. Measurable disease at time of enrollment according to the revised international working group response criteria for malignant lymphoma.
5. Life expectancy ≥12 weeks
6. Eastern Cooperative Oncology Group (ECOG) performance status that is either 0 or 1 at screening.
7. Adequate organ function:

   * Renal function defined as:

     * A serum creatinine of ≤1.5 x Upper Limit of Normal(ULN) or
     * Estimated Glomerular Filtration Rate (eGFR) ≥ 60 mL/min/1.73 m2
   * Liver function defined as:

     * Alanine Aminotransferase (ALT) ≤ 5 times the ULN for age
     * Bilirubin ≤ 2.0 mg/dl with the exception of patients with Gilbert-Meulengracht syndrome; patients with Gilbert-Meulengracht syndrome may be included if their total bilirubin is ≤ 3.0 x ULN and direct bilirubin ≤ 1.5 x ULN
   * Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and pulse oxygenation > 91% on room air
8. Hemodynamically stable and Left Ventricle Ejection Fraction (LVEF) ≥ 45% confirmed by echocardiogram or Multigated Radionuclide Angiography (MUGA)
9. Adequate bone marrow reserve without transfusions defined as:

   * Absolute neutrophil count (ANC) > 1000/μL
   * Absolute lymphocyte count (ALC) ≥ 300/μL
   * Platelets ≥ 50000/μL
   * Hemoglobin > 8.0 g/dl
10. Must have an apheresis product of non-mobilized cells accepted for manufacturing.
11. The following medications are excluded:

    * Steroids: Therapeutic doses of steroids must be stopped > 72 hours prior to BZ019 infusion. However, the following physiological replacement doses of steroids are allowed: < 6 - 12 mg/m2/day hydrocortisone or equivalent
    * Immunosuppression: Any immunosuppressive medication must be stopped ≥ 4 weeks prior to enrollment
    * Antiproliferative therapies other than lymphodepleting chemotherapy within two weeks of infusion
    * Antibody use including anti-CD20 therapy within 4 weeks prior to infusion or 5 half-lives of the respected antibody, whichever is longer
    * CNS disease prophylaxis must be stopped > 1 week prior to BZ019 infusion (e.g. intrathecal methotrexate)
12. Women of child-bearing potential (defined as all women physiologically capable of becoming pregnant) and all male participants must agree to use highly effective methods of contraception for at least 12 months following BZ019 infusion and until CAR T cells are no longer present by PCR on two consecutive tests

Exclusion Criteria:

1. Prior treatment with any prior anti-CD19/anti-CD3 therapy, or any other anti-CD19 therapy
2. Treatment with any prior gene therapy product, include CAR-T cell therapy.
3. Active Central Nervous System (CNS) involvement by malignancy or secondary CNS involvement
4. History or presence of clinically relevant CNS pathology such as epilepsy, seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or self-immune disease with CNS involvement.
5. Prior allogeneic HSCT
6. Eligible for and consenting to ASCT
7. Chemotherapy other than lymphodepleting chemotherapy within 2 weeks of infusion
8. Investigational medicinal product within the last 30 days prior to screening
9. Prior radiation therapy within 2 weeks of infusion
10. Active replication of or prior infection with hepatitis B or active hepatitis C( HCV RNA positive )
11. HIV positive patients
12. Uncontrolled acute life threatening bacterial, viral or fungal infection (e.g. blood culture positive ≤ 72 hours prior to infusion)
13. Unstable angina and/or myocardial infarction within 6 months prior to screening
14. Previous or concurrent malignancy with the following exceptions:

    * Adequately treated basal cell or squamous cell carcinoma (adequate wound healing is required prior to study entry)
    * In situ carcinoma of the cervix or breast, treated curatively and without evidence of recurrence for at least 3 years prior to the study
    * A primary malignancy which has been completely resected and in complete remission for ≥ 5 years
15. Pregnant or nursing (lactating) women
16. Cardiac arrhythmia not controlled with medical management
17. Patients on oral anticoagulation therapy within 1 week prior to BZ019 infusion.
18. Prior treatment with any adoptive T cell therapy
19. Patients with active neurological auto immune or inflammatory disorders(e.g. Guillain Barre Syndrome, Amyotrophic Lateral Sclerosis)
20. Other protocol-related inclusion/exclusion may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | up to 1 year after BZ019 infusion.
  Number of BZ019 therapy associated adverse events, such as cytokine release syndrome(CRS), chimeric antigen receptor (CAR)-T cell related encephalopathy syndrome(CRES) or other adverse events.

SECONDARY OUTCOMES:
proliferation of BZ019 in vivo | up to 1 year after BZ019 infusion.
  measured by PCR
Overall response rate | up to 1 year after BZ019 infusion.
  CR+PR

CONTACTS AND LOCATIONS:
Overall Officials: Lugui Qiu, MD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No